CLINICAL TRIAL: NCT03641196
Title: Bonded, Cemented or Removable Orthodontic Approaches to Correct Deep Bite in Mixed Dentition Patients: a Randomized Controlled Trial
Brief Title: Orthodontic Approaches to Correct Deep Bite in Mixed Dentition Patients
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The study was terminated due to difficulties in the recruitment attributed to the Covid19 pandemic.
Sponsor: University of Alberta (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Pro00082429
Record Dates: First submitted 2018-08-14; First posted 2018-08-21 (Actual); Last update posted 2022-05-23 (Actual); Status verified 2019-10

CONDITIONS: Overbite (Excessive) Deep
Keywords: Orthodontic Appliances; Dentition, Mixed
MeSH Terms: conditions — Overbite | interventions — Orthodontic Appliances, Fixed

STUDY DESIGN:
Intervention Model Description: This study will be a stratified, parallel randomized controlled, single-blinded, with an allocation ratio of 1:1:1.
Who Masked: Outcomes Assessor
Masking Description: The analyses will be blinded regarding treatment received and time.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- No treatment of deep bite (No Intervention): No treatment of deep bite. These participants will be evaluated during a 6-month follow-up period. In cases were significant problems arise during the follow-up period, the participant will be removed from the study and the appropriate treatment conducted.
- Fixed appliance (Active Comparator): Fixed appliance: Treatment with a cemented modified palatal Nance appliance presenting a bite-plane.
  Interventions: Device: Fixed appliance
- Composite bite plane (Active Comparator): Composite bite plane: Treatment with a composite build up in the palatal aspect of the upper central incisors.
  Interventions: Procedure: Composite bite plane

INTERVENTIONS:
Device: Fixed appliance — Use of a cemented modified palatal Nance appliance presenting a bite-plane
  Arms: Fixed appliance
Procedure: Composite bite plane — treatment with a composite build up in the palatal aspect of the upper central incisors.
  Arms: Composite bite plane

SUMMARY:
A deep bite is a bite where the upper front teeth cover almost all, if not all the lower front teeth.

Currently there is no clarity which of the available treatment approaches is better when these patients still have some baby (deciduous) teeth in their mouths.

This study will compare the results of four ways to manage this problem:

1. Delay treatment until all permanent teeth are erupted,
2. Temporary glue some brackets to the upper front teeth and correct the problem with orthodontic wires,
3. Temporary glue some dental material in the back of the front teeth to allow the back teeth to erupt.

The amount of improvement (increased exposure of lower front teeth when biting) will be compared between the four treatment options.

The reason there is a no treatment group is because a slight improvement of the deep bite happens naturally in some cases. In this case delay of treatment is not a major concern as this bite type can be managed later during permanent dentition.

DETAILED DESCRIPTION:
Purpose: Deep bite, an increase from the normal overbite, is a problem that can be caused by a dentoalveolar and/or skeletal origin, and it is more common in class II malocclusion patients. Among children, the prevalence has been reported to range from 3 to 39%. This large variance can be explained by factors such as diagnosis criteria, sex, and ethnic group. Even though the stability and relapse of deep bite treatment have been previously discussed on permanent dentition, there is a lack of studies investigating their management during mixed dentition. Hence the goal of this clinical trial is to assess if any of the currently available approaches is more efficient considering factors such as costs, number of appointments, complications and patient's experience.

Hypothesis: The investigators hypothesized that the three active treatment approaches (bonded vs. cemented vs. removable) would produce similar dentoalveolar, skeletal and functional improvements. Those improvements would be larger than those observed on untreated children.

Justification: There is a lack of evidence regarding what early treatment approach for the deep bite is more effective, produces fewer side effects, and is more comfortable for patients. No randomized controlled trial evaluating the effectiveness of deep bite treatment during the mixed dentition has been identified. Early intervention may simplify future comprehensive orthodontic treatment. Moderate to severe deep bite cases could affect sagittal mandibular growth.

Objectives: This study aims to evaluate the effectiveness of two deep bite orthodontic treatments among children in the mixed dentition phase. Additionally, treatment duration, quality of life changes and complications of the different performed interventions will be assessed.

Research Method/Procedures: This study will be a stratified, parallel randomized controlled, single-blinded, with an allocation ratio of 1:1:1. The sample will be composed by children in mixed dentition (7-11 year olds), referred or self-referred to the orthodontic clinic at the University of Alberta (Edmonton, Alberta, Canada). The inclusion criteria will be: presence of moderate to severe deep bite (overbite >5.0 mm), fully erupted maxillary and mandibular incisors, as well as first permanent molars, no missing permanent incisors and molars, no clinically noticeable craniofacial syndromes and no clear need for immediate intervention to manage severe sagittal, transversal or vertical malocclusions. The participants will be divided into three groups:

1. no treatment of deep bite now - deferral to permanent dentition;
2. treatment with a cemented modified palatal Nance appliance including an anterior bite-plane;
3. treatment with a composite build up in the palatal aspect of the upper central incisors.

The effectiveness of interventions (elimination of the moderate to severe anterior deep bite) will be assessed as a primary outcome. Secondarily, treatment duration, compliance, and complications among patients using the appliances will be evaluated. The treatment effectiveness will be evaluated according to the following criteria:

* The success rate of deep overbite correction (yes or no). The success in overbite correction will be defined as the complete dissolution of deep bite, with an overbite <3mm. This will be assessed by comparing digital bite models from before (T0) and after treatment (T1).
* Treatment duration in months: from the beginning until the end of the intervention (correction of deep bite up to a maximum of 12 months). The number of appointments will also be calculated.
* Measurement of overjet and overbite in millimeters; arch length to incisal edge in millimeters; maxillary dental arch length total (ALT) in millimeters; transverse maxillary molar distance (MD) in millimeters. Obtained from digital bite models.
* Cephalometric analysis. Skeletal and vertical sagittal measurements, as well as interdental, maxillary and mandibular dentoalveolar measurements, will be collected for each participant. Conventional 2-D Lateral cephalograms will be taken from all patients before treatment (T0) and at the end of the active intervention (T1).

The overjet, overbite, and the arch length will be measured electronically. Cephalometric measurements will be made with a commercial software. All measurements were made to the nearest 0.1 mm by an orthodontist. The analyses will be blinded regarding treatment received and time. Changes in the different measures were calculated as the difference between T1 and T0. Finally, the duration of treatment (no more than 12 months) will be considered.

Data on all patients will be analyzed on an intention-to-treat (ITT) basis, i.e., if the deep bite was not corrected during the 1-year trial period, the outcome will be declared unsuccessful. Thus, all patients, successful or not, will be included in the final analysis. The dropouts during the trial will be evaluated regarding the reasons and the data collected during the study to be considered as effective or ineffective.

Cephalometric and digital bite models measurements of 10 patients will be repeated by the same observer, a trained orthodontist, after four weeks to measure the intraobserver reliability. The reliability will be measured using Dahlberg formula for random error analysis and intraclass correlation (ICC) for the evaluation of systematic errors.

As a secondary outcome, the number of breakages, additional appointments for appliance repairs, appliance repairs made and emergency appointments will be collected to evaluate the complications of each treatment. In the removable appliance group, the compliance will be evaluated using a using an incorporated microsensor.

Quality of life will be assessed using previously validated questionnaires specific to age groups. For 8 to 10 year-old the CPQ8-10 which consists of 25 questions distributed among 4 domains (oral symptoms, functional limitations, emotional well-being and social well-being). For 11 to 12-year-old the CPQ11-14 which consists of 37 questions distributed among 4 domains (oral symptoms, functional limitations, emotional well-being and social well-being). The P-CPQ, a measure of parental/caregiver perceptions of the oral health-related quality of life of children will also be used.

The sample size was calculated based on a power analysis, considering overbite as the primary variable. To achieve a power of the study of 0.8, a difference among treatments of 1mm (variance of 1.5mm2) at a level of 0.05, each group of patients under investigation had to include 24 subjects. Considering a possible dropout rate of 20% in each group, 29 subjects will be recruited in each group, resulting in a total initial sample of 87 children. Data from Bacetti et al 2012 study comparing deep bite correction between mixed mention and permanent dentition used as reference (1.7 mm difference with sd of 1.3 mm).

A computer-generated list of random numbers will be used to randomly selected sample from a large pool of participants (SPSS Inc., Chicago.). This process will be conducted by a person not involved in the study. The random allocation process will be performed using opaque sealed envelopes which will contain the assigned group for each patient and were not opened until the onset of the trial. The enrolment of participants and their assignment will be done by an orthodontic staff member not directly involved in the intervention and follow-up. A computer-generated list of random numbers will be used to randomly selected sample from a large pool of participants (SPSS Inc., Chicago.). This process will be conducted by a person not involved in the study. The random allocation process will be performed using opaque sealed envelopes which contained the assigned group for each patient and were not opened until the onset of the trial.

Plan for Data Analysis: Data normality will be examined using the Shapiro-Wilk test. A multiple analysis of variance (MANOVA) will be used to evaluate repeated-measures data between T0 and T1 in each group. Intergroup comparison among different intervention groups will be performed using multiple analyses of variance (MANOVA), with Tukey ́s posthoc test. All statistical analyses will be conducted using IBM SPSS Statistics 22 (SPSS Inc., Chicago, IL, USA) software, with a 0.05 level of significance.

ELIGIBILITY:
Inclusion Criteria:

* presence of moderate to severe deep bite (overbite, >5.0 mm);
* fully erupted maxillary and mandibular incisors, as well as first permanent molars.

Exclusion Criteria:

* missing permanent incisors and molars;
* clinically noticeable craniofacial syndromes;
* need for immediate intervention to assess severe sagittal, transversal or vertical malocclusions.

Min Age: 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2019-01-15 (Actual); Primary Completion 2021-09-10 (Actual); Study Completion 2021-09-10 (Actual)

PRIMARY OUTCOMES:
Elimination of the moderate to severe anterior deep bite | The success rate was assessed by comparing study models from before (T0) and after treatment (T1)(no more than 12 months).
  The success in overbite correction (yes/no) will be defined as the complete dissolution of deep bite, with an overbite 3mm.
Measurement of overjet and overbite | Before (T0) and after treatment (T1) (no more than 12 months).
  Measurement of overjet and overbite in millimeters, using a measured with a pencil and ruler. All measurements were made to the nearest 0.1 mm by an orthodontist.Obtained from digital bite models.
Arch length to incised edge | Before (T0) and after treatment (T1) (no more than 12 months).
  Measurement of the arch length to incisal edge, in millimeters, using a measured with a pencil and ruler. All measurements were made to the nearest 0.1 mm by an orthodontist. Obtained from digital bite models.
Maxillary dental arch length total | Before (T0) and after treatment (T1) (no more than 12 months).
  Measurement of the total maxillary dental arch length, in millimeters, using a measured with a pencil and ruler. All measurements were made to the nearest 0.1 mm by an orthodontist. Obtained from digital bite models.
Transverse maxillary molar distance | Before (T0) and after treatment (T1) (no more than 12 months).
  Measurement of the transverse maxillary molar distance, in millimeters, using a measured with a pencil and ruler. All measurements were made to the nearest 0.1 mm by an orthodontist. Obtained from digital bite models.
Cephalometric analysis | Before (T0) and after treatment (T1) (no more than 12 months).
  Cephalometric measures, including sagittal interdental, maxillary and mandibular dentoalveolar measurements, will be collected for each participant. All these measurements will be combined on a final evaluation of craniofacial changes. Conventional 2-D Lateral cephalograms will be taken from all patients before treatment (T0) and at the end of the active intervention (T1). A trained and calibrated orthodontist, previously calibrated will perform the measurements.

SECONDARY OUTCOMES:
Treatment duration in months | correction of deep bite up to a maximum of 12 months
  from the beginning until the end of the intervention
Breakages | 12 months
  The number of breakages will be recorded during the follow-up period.
Additional appointments | 12 months
  The number of additional appointments for appliance repairs will be recorded during the follow-up period.
Emergency appointments | 12 months
  The number of emergency appointments will be recorded during the follow-up period.
Compliance in the removable appliance group | 12 months
  The compliance will be evaluated using a using an incorporated microsensor.
Quality of life measurement | Before (T0) and after treatment (T1) (no more than 12 months).
  Quality of life will be assessed using previously validated questionnaires specific for age groups. For 8 to 10 year-old the CPQ8-10 which consists of 25 questions distributed among 4 domains (oral symptoms, functional limitations, emotional well-being and social well-being). For 11 to 12 year-old the CPQ11-14 which consists of 37 questions distributed among 4 domains (oral symptoms, functional limitations, emotional well-being and social well-being). The P-CPQ, a measure of parental/caregiver perceptions of the oral health-related quality of life of children will also be used.

CONTACTS AND LOCATIONS:
Overall Officials: Carlos Flores-Mir, PhD, Principal Investigator — University of Alberta
Locations (1):
- Orthodontic clinic at the University of Alberta, Edmonton, Alberta, Canada

IPD SHARING:
Plan to Share IPD: Undecided
The sharing of individual participant data was not yet decided.

REFERENCES:
- [Background] Huang GJ, Bates SB, Ehlert AA, Whiting DP, Chen SS, Bollen AM. Stability of deep-bite correction: A systematic review. J World Fed Orthod. 2012 Sep 1;1(3):e89-e86. doi: 10.1016/j.ejwf.2012.09.001. PMID 23630651
- [Background] Feldmann I, Lundstrom F, Peck S. Occlusal changes from adolescence to adulthood in untreated patients with Class II Division 1 deepbite malocclusion. Angle Orthod. 1999 Feb;69(1):33-8. doi: 10.1043/0003-3219(1999)0692.3.CO;2. PMID 10022182
- [Background] de Souza BS, Bichara LM, Guerreiro JF, Quintao CC, Normando D. Occlusal and facial features in Amazon indigenous: An insight into the role of genetics and environment in the etiology dental malocclusion. Arch Oral Biol. 2015 Sep;60(9):1177-86. doi: 10.1016/j.archoralbio.2015.04.007. Epub 2015 May 21. PMID 26051559
- [Background] Ferro R, Besostri A, Olivieri A, Stellini E. Prevalence of occlusal traits and orthodontic treatment need in 14 year-old adolescents in Northeast Italy. Eur J Paediatr Dent. 2016 Mar;17(1):36-42. PMID 26949237
- [Background] Lux CJ, Ducker B, Pritsch M, Komposch G, Niekusch U. Occlusal status and prevalence of occlusal malocclusion traits among 9-year-old schoolchildren. Eur J Orthod. 2009 Jun;31(3):294-9. doi: 10.1093/ejo/cjn116. Epub 2009 Feb 25. PMID 19244457
- [Background] Silness J, Roynstrand T. Effects of the degree of overbite and overjet on dental health. J Clin Periodontol. 1985 May;12(5):389-98. doi: 10.1111/j.1600-051x.1985.tb00929.x. PMID 3859497
- [Background] Bergersen EO. A longitudinal study of anterior vertical overbite from eight to twenty years of age. Angle Orthod. 1988 Jul;58(3):237-56. doi: 10.1043/0003-3219(1988)0582.0.CO;2. PMID 3189955
- [Background] Grippaudo C, Pantanali F, Paolantonio EG, Saulle R, Latorre G, Deli R. Orthodontic treatment timing in growing patients. Eur J Paediatr Dent. 2013 Sep;14(3):231-6. PMID 24295010
- [Background] Baccetti T, Franchi L, Giuntini V, Masucci C, Vangelisti A, Defraia E. Early vs late orthodontic treatment of deepbite: a prospective clinical trial in growing subjects. Am J Orthod Dentofacial Orthop. 2012 Jul;142(1):75-82. doi: 10.1016/j.ajodo.2012.02.024. PMID 22748993
- [Background] Hellsing E. Increased overbite and craniomandibular disorders--a clinical approach. Am J Orthod Dentofacial Orthop. 1990 Dec;98(6):516-22. doi: 10.1016/0889-5406(90)70018-8. PMID 2248230
- [Background] Franchi L, Baccetti T, Giuntini V, Masucci C, Vangelisti A, Defraia E. Outcomes of two-phase orthodontic treatment of deepbite malocclusions. Angle Orthod. 2011 Nov;81(6):945-52. doi: 10.2319/033011-229.1. Epub 2011 Jul 29. PMID 21801005
- [Background] Baccetti T, Franchi L, McNamara JA Jr. Longitudinal growth changes in subjects with deepbite. Am J Orthod Dentofacial Orthop. 2011 Aug;140(2):202-9. doi: 10.1016/j.ajodo.2011.04.015. PMID 21803258